CLINICAL TRIAL: NCT03445702
Title: Metformin Gastrointestinal Intolerance: Measurement of Mitochondrial Complex I
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Alexis McKee, MD, MD, St. Louis University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: 25319
Record Dates: First submitted 2018-02-19; First posted 2018-02-26 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2; Metformin Adverse Reaction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Randomized, double blinded, placebo controlled crossover trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigators, participants, research coordinator will be blinded to intervention provided to subject
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Metformin intolerant & metformin (Experimental): Metformin 1000mg once
  Interventions: Drug: Metformin
- Metformin intolerant & placebo (Placebo Comparator): Placebo 1000mg once
  Interventions: Drug: Placebo
- Metformin tolerant & metformin (Active Comparator): Metformin 1000mg once
  Interventions: Drug: Metformin
- Metformin tolerant and placebo (Placebo Comparator): Placebo 1000mg once
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1000mg once
  Other Names: Glucophage
  Arms: Metformin intolerant & metformin; Metformin tolerant & metformin
Drug: Placebo — Sugar pill manufactured to mimic metformin 1000mg
  Arms: Metformin intolerant & placebo; Metformin tolerant and placebo

SUMMARY:
Metformin is associated with a high degree of gastrointestinal intolerance, which limits the effective use of the medication. It is proposed to be an inhibitor of liver mitochondrial glycerophosphate dehydrogenase which results in partial blockade of mitochondrial complex 1 and inhibition of metabolism of lactate to pyruvate. There is also evidence that it is accumulated in gastrointestinal cells, and that there are certain genotypes associated with inclusion or lack of exclusion of the metformin from these cells. To validate this hypothesis investigators propose to give metformin after a standard meal test to see if there is the accumulation of lactic acid in those with gastrointestinal intolerance to metformin, compared to those without intolerance, and to determine if these elevations of lactic acid and GI symptoms are associated with genetic predispositions.

Aims:

1. To determine if the GI intolerance to metformin is associated with post meal elevations of lactic acid.

   a. The test will measure the inhibition of mitochondrial complex 1 levels of lactate to pyruvate compared with non- intolerant subjects.
2. To determine if individuals with gastrointestinal symptoms and elevated lactate/pyruvate ratios have genetic variation in the organic cation transporters.

DETAILED DESCRIPTION:
Metformin is the primary drug of choice for management of type 2 diabetes mellitus. Most recent evidence suggest that the drug is a noncompetitive inhibitor of mitochondrial glycerophosphate dehydrogenase which modifies mitochondrial complex 1 in the liver, reducing the generation of NADH, increasing the ratio of lactate to pyruvate, and reducing gluconeogenesis. Metformin which is a guanidine/ biguanide analog is not metabolized in vivo and is cleared by the kidney. It has a limited degree of mitochondrial inhibition, and only becomes toxic when serum levels accumulate in renal failure. Other guanidine analogs, such as fenformin or galegine, however may be associated with irreversible complete mitochondrial blockade and lactic acidosis.

The incidence of gastrointestinal intolerance to the drug can range between 10% and 30%. It is postulated that the gastrointestinal enterocyte may accumulate the metformin. It is postulated that metformin uptake and accumulation may be exacerbated in those with genetic predispositions for certain organic transporters which are involved in the uptake and removal of metformin in cells. Metformin appears to be taken up from the intestine by plasma monoamine transporter (PMAT; SLC29A4), organic cation transporter 1 (OCT1; SCLC22A1) and organic cation transporter 3 (OCT3; SLC22A3) and actively removed from target tissues by multi-antimicrobial extrusion protein 1 (MATE1; SLC47A1) and eliminated by the urinary multi-antimicrobial extrusion protein 2 (MATE2; SCL47A2). Although certain genotypes are associated with a high incidence of intolerance, the gene low gene frequency does not explain the high degree of intolerance in the population.

ii) Innovation: The plan is to develop a test to evaluate whether there is accumulation of lactic acid after a therapeutic dose of metformin and whether the levels of lactic acid are higher in subjects with GI intolerance than those not intolerant. The hypothesis is that there is increased generation of lactic acid in those intolerant individuals, independent of glucose lowering effect on liver metabolism. Investigators propose to measure the generation of lactate/pyruvate (L/P, mitochondrial complex 1), in those with and without clinically known metformin gastrointestinal symptoms. Investigators will correlate gastrointestinal symptoms with L/P ratios. Investigators will also evaluate for genomic susceptibility for the origin transporters with comparison to the metformin tolerance test generation of lactic acid.

iii) Approach: Investigators wish to develop a pilot project of 24 subjects who will complete the protocol. Subject will be seen in the Endocrinology clinic of St. Louis University, and investigators will recruit 12 subjects who have clinical symptoms of gastrointestinal symptoms (diarrhea or bloating) and 12 subjects who are tolerant. Subjects will be randomized to receive a fasting standard dose of 1000 mg brand metformin (Glucophage) or comparable placebo on day one and then the alternate medicine on a second day. The study drug will be given with Diabetasourse meal (standard meal) which will provide carbohydrates to challenge the mitochondrial system [2]. Bloods for glucose, L/P, will be obtained at 0, 30 60 90 and 120 minutes. Symptoms of gastrointestinal effects will be documented by a Likert type questionnaire. Outcomes will be 1) the effect of metformin vs. placebo on the meal tolerance glucose levels 2) the effect of metformin on post meal challenge levels of L/P, in intolerant vs. tolerant individual and 3) the correlation of gastrointestinal symptoms with changes in L/P. From animal data, metformin causes a 2 fold increase in lactic acid at 60 minutes. In our laboratory with a normal reference lactic acid of 1.0 mmol/L and a SD=0.725. Twelve pairs would be sufficient for a pilot study to determine a difference at an alpha of 0.05 and beta of 0.80.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus
2. Tolerance to meformin
3. Intolerance to metformin

Exclusion Criteria:

1. Exclusion: Pregnant or nursing mothers
2. Those not competent to provide informed consent
3. Known systemic allergy (not intolerance) to metformin
4. Congestive heart failure NYHA class III-IV
5. Renal impairment,EGFRr<45ml/min
6. Liver cirrhosis

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2020-10-27 (Actual)

PRIMARY OUTCOMES:
Lactate to pyruvate ratio | 2 weeks
  Meal tolerance test. Absolute levels and ratios of L/P will be compared pre and post metformin and between group by analysis of variance for repeated measures where the covariance is group (tolerant or intolerant) and drug (metformin vs placebo).

SECONDARY OUTCOMES:
Genomic testing | 2 weeks
  The subjects will have genomic testing for variations in cellular transporters

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ferrannini E. The target of metformin in type 2 diabetes. N Engl J Med. 2014 Oct 16;371(16):1547-8. doi: 10.1056/NEJMcibr1409796. No abstract available. PMID 25317875
- [Background] Madiraju AK, Erion DM, Rahimi Y, Zhang XM, Braddock DT, Albright RA, Prigaro BJ, Wood JL, Bhanot S, MacDonald MJ, Jurczak MJ, Camporez JP, Lee HY, Cline GW, Samuel VT, Kibbey RG, Shulman GI. Metformin suppresses gluconeogenesis by inhibiting mitochondrial glycerophosphate dehydrogenase. Nature. 2014 Jun 26;510(7506):542-6. doi: 10.1038/nature13270. Epub 2014 May 21. PMID 24847880
- [Background] Bailey CJ, Wilcock C, Scarpello JH. Metformin and the intestine. Diabetologia. 2008 Aug;51(8):1552-3. doi: 10.1007/s00125-008-1053-5. Epub 2008 Jun 5. No abstract available. PMID 18528677
- [Background] Bailey CJ, Wilcock C, Day C. Effect of metformin on glucose metabolism in the splanchnic bed. Br J Pharmacol. 1992 Apr;105(4):1009-13. doi: 10.1111/j.1476-5381.1992.tb09093.x. PMID 1504710
- [Background] Buse JB, DeFronzo RA, Rosenstock J, Kim T, Burns C, Skare S, Baron A, Fineman M. The Primary Glucose-Lowering Effect of Metformin Resides in the Gut, Not the Circulation: Results From Short-term Pharmacokinetic and 12-Week Dose-Ranging Studies. Diabetes Care. 2016 Feb;39(2):198-205. doi: 10.2337/dc15-0488. Epub 2015 Aug 18. PMID 26285584
- [Background] Tarasova L, Kalnina I, Geldnere K, Bumbure A, Ritenberga R, Nikitina-Zake L, Fridmanis D, Vaivade I, Pirags V, Klovins J. Association of genetic variation in the organic cation transporters OCT1, OCT2 and multidrug and toxin extrusion 1 transporter protein genes with the gastrointestinal side effects and lower BMI in metformin-treated type 2 diabetes patients. Pharmacogenet Genomics. 2012 Sep;22(9):659-66. doi: 10.1097/FPC.0b013e3283561666. PMID 22735389
- [Background] Pawlyk AC, Giacomini KM, McKeon C, Shuldiner AR, Florez JC. Metformin pharmacogenomics: current status and future directions. Diabetes. 2014 Aug;63(8):2590-9. doi: 10.2337/db13-1367. PMID 25060887
- [Background] Wang L, Weinshilboum R. Metformin pharmacogenomics: biomarkers to mechanisms. Diabetes. 2014 Aug;63(8):2609-10. doi: 10.2337/db14-0609. No abstract available. PMID 25060891
- [Background] Davidson J, Howlett H. New prolonged-release metformin improves gastrointestinal tolerability. British Journal of Diabetes & Vascular Disease 2004; 4: 273.
- [Background] Blonde L, Dailey GE, Jabbour SA, Reasner CA, Mills DJ. Gastrointestinal tolerability of extended-release metformin tablets compared to immediate-release metformin tablets: results of a retrospective cohort study. Curr Med Res Opin. 2004 Apr;20(4):565-72. doi: 10.1185/030079904125003278. PMID 15119994